CLINICAL TRIAL: NCT06577259
Title: A Phase 1, Open-label, Single-site, Randomized, Single-dose, Three-way, Crossover Study to Assess the Relative Bioavailability of BMS-986435 Tablet Formulations in Healthy Adult Participants
Brief Title: Study to Assess Relative Bioavailability of BMS-986435 Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV029-1018
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: BMS-986435; MYK-224; Healthy participants; Single-dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: BMS-986435 Reference Dose 1 (Active Comparator)
  Interventions: Drug: BMS-986435
- Treatment B: BMS-986435 Test Dose 1 (Experimental)
  Interventions: Drug: BMS-986435
- Treatment C: BMS-986435 Test Dose 2 (Experimental)
  Interventions: Drug: BMS-986435

INTERVENTIONS:
Drug: BMS-986435 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the relative bioavailability of BMS-986435 tablet formulations in healthy adult male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 45 kg and a body mass index (BMI) between 18 and 32 kg/m^2, inclusive.
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) and clinical laboratory assessments.
* Have documented left ventricular ejection fraction (LVEF) ≥ 60% and absence of significant cardiac abnormality.

Exclusion Criteria:

* Any acute or chronic medical illness.
* History of heart disease.
* Prior exposure to BMS-986435.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 105 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration [AUC(0-T)] | Up to 105 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | Up to 105 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve truncated at 72 hour [AUC(0-72h)] | Up to 105 days
Time of maximum observed concentration [Tmax] | Up to 105 days
Apparent terminal half-life [T-HALF] | Up to 105 days
Incidence of adverse events (AEs) | Up to approximately 5 months
Incidence of serious adverse events (SAEs) | Up to approximately 5 months
Incidence of participants with vital sign abnormalities | Up to 105 days
Incidence of participants with physical examinations abnormalities | Up to 105 days
Incidence of participants with electrocardiogram (ECG) abnormalities | Up to 105 days
Incidence of participants with clinical laboratory abnormalities | Up to 105 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com